CLINICAL TRIAL: NCT06329388
Title: A Six-Month Randomized Controlled Pilot Study Evaluating the Effects of an Oral Protein Supplement on Children's Growth Patterns
Brief Title: Evaluating the Effects of an Oral Protein Supplement on Children's Growth Patterns
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TruHeight Vitamins (Industry)
Collaborators: San Francisco Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSD-SFRI-013
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Growth Disorders; Dietary Exposure; Child Development; Bone Development Abnormal; Body Weight; Child Malnutrition
Keywords: Children's Growth Patterns; Oral Protein Supplement; Pediatric Nutrition; Growth Supplements; Height Increase; Type X Collagen; Body Composition Analysis; Dietary Intervention; Nutritional Status in Children; Randomized Controlled Trial (RCT); Child Development; INBODY Device; Safety and Tolerability of Protein Shakes; Bone Growth Markers; Nutritional Supplements and Child Growth; TruHeight
MeSH Terms: conditions — Growth Disorders; Body Weight; Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT) with two parallel groups (treatment and control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment - Oral Protein Supplement (Experimental): Participants in this arm will receive the TruHeight Growth Protein Shake. Each serving consists of two scoops of the supplement powder mixed with 12-16 fluid ounces of water. The regimen is once daily, five times per week, for a duration of six months.
  Interventions: Dietary Supplement: TruHeight Growth Protein Shake
- Control - No Supplement (No Intervention): Participants in this arm will not receive the oral protein supplement but will continue their regular diet. They serve as a comparison group to evaluate the effects of the TruHeight Growth Protein Shake administered to the treatment group.

INTERVENTIONS:
Dietary Supplement: TruHeight Growth Protein Shake — Participants will be administered two scoops of TruHeight Growth Protein Shake, mixed with 12-16 fluid ounces of water, once daily, five times per week for six months. The supplement is intended to support growth patterns in children by providing essential nutrients that contribute to bone development and overall growth.
  Arms: Treatment - Oral Protein Supplement

SUMMARY:
This single-center, randomized controlled pilot study aims to evaluate the efficacy of TruHeight Growth Protein Shake on improving growth patterns in children aged 4-17 years. Over six months, participants will consume the protein shake daily, five times a week, with outcomes measured in terms of type X collagen concentration in urine, height via a stadiometer, and body composition using an INBODY device.

DETAILED DESCRIPTION:
This single-center pilot clinical trial was conducted for TruHeight to determine the effect of oral protein supplement (Growth Protein Shake-GPS) versus control on growth patterns in children. The hypothesis posits that GPS protein supplementation will improve growth patterns as assessed by the concentration of collagen X in the urine, height as measured by a stadiometer, as well as weight and body composition as measured by an INBODY device in six months.

The oral supplement was provided in powder form, which could be mixed with water before consumption.

Participants were recruited from the SF RESEARCH INSTITUTE database and through advertisements on social media and public places. Initial attendance at SF RESEARCH INSTITUTE marked the baseline study visit, where subjects underwent screening for eligibility based on the Inclusion and Exclusion Criteria. Upon meeting qualification criteria, enrollees were assigned a subject number sequentially as they joined the study. A total of 32 subjects, aged 4-17 years, embarked on the study, targeting a completion cohort of 20. Randomization into either the treatment/supplement group or control group occurred via a computer-generated code.

The trial comprised three study visits (SV) over a 6-month period. Measurements of height, weight, fat mass, and lean body mass took place at baseline (SV1), 3 months ± 5 days (SV2), and 6 months ± 5 days (SV3). Urine samples collected at SV1 and SV3 underwent laboratory analysis for type X collagen content. Depending on the group assignment, a dietary or consumer perception questionnaire was provided to be completed by the participant or the participant's guardian at baseline, SV2, and SV3. Treatment group participants or their guardians received a log form to document supplement intake at home. Maintenance of regular diet throughout the study was mandatory for all participants.

Instructions for subjects in the treatment/supplement group were as follows:

Mix and consume two (2) scoops of the dietary supplement with 12-16 fluid oz of water daily, five times per week, for 6 months. The investigator initiated follow-up calls to subjects or their guardians on day 45 (between SV1 and SV2) and day 120 (between SV2 and SV3) to assess compliance with the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-17 years old
* At or below the 50th percentile for height according to CDC growth charts
* Able to consume the protein shake
* Willing to maintain their regular diet throughout the study

Exclusion Criteria:

* Known allergies to ingredients in the protein shake
* Currently receiving growth hormone therapy
* Any medical condition that can affect growth or requires special diet

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Change in Height | 6 months
  The primary measure is the difference in children's height measured by a stadiometer from baseline to the end of the study at six months.

SECONDARY OUTCOMES:
Change in Type X Collagen Concentration in Urine | Baseline and 6 months
  Measure the difference in Type X collagen concentration in urine samples from baseline to the end of the study to assess bone growth.
Change in Body Composition | Baseline, 3 months, and 6 months
  Evaluate the difference in body composition, including fat mass and lean body mass percentage, using the INBODY device from baseline to the end of the study.
Incidence of Adverse Events | Throughout the study period of 6 months
  Monitor and record any adverse events experienced by participants throughout the study duration.

CONTACTS AND LOCATIONS:
Locations (1):
- SF Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The study proposes to share individual participant data that underlie the results reported in an article after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Starting at 6 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal for use of the data in a peer-reviewed publication may access the data.
URL: https://truheightvitamins.com/pages/clinical-study

REFERENCES:
- See also: Wikipedia contributors. (2023). Stadiometer. In Wikipedia — https://en.wikipedia.org/wiki/Stadiometer
- See also: Innovative Research. (n.d.). Human Collagen Type X ELISA Kit — https://www.innov-research.com/products/human-collagen-type-x-elisa-kit
- See also: Gudmann, N., & Karsdal, M. (2016). Type X Collagen. In Elsevier eBooks (pp. 73-76) — https://doi.org/10.1016/b978-0-12-809847-9.00010-6
- See also: Voss, L. D., Bailey, B. J., Cumming, K., Wilkin, T. J., & Betts, P. R. (1990). The reliability of height measurement (the Wessex Growth Study). Archives of Disease in Childhood, 65(12), 1340-1344 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC1792390/
- See also: Voss, L. D., & Wilkin, T. J. (1991). The reliability of height and height velocity in the assessment of growth (the Wessex Growth Study). Archives of Disease in Childhood, 66(8), 833-837 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC1793253/
- See also: Van den Broeck, J., Hokken-Koelega, A., & Wit, J. (1999). Validity of height velocity as a diagnostic criterion for idiopathic growth hormone deficiency and Turner syndrome. Hormone Research, 51(2), 68-73 — https://www.pubmed.ncbi.nlm.nih.gov/10352397/
- See also: Linsenmayer, T. F., Eavey, R. D., & Schmid, T. M. (1988). Type X collagen: A hypertrophic cartilage-specific molecule. Pathology and Immunopathology Research, 7(1), 14-19 — https://www.pubmed.ncbi.nlm.nih.gov/3283937/
- Available data/document: Clinical Study Report — https://www.truheightvitamins.com/pages/clinical-study — Submit your email to have a copy of the Clinical Trial sent to you.